CLINICAL TRIAL: NCT04768803
Title: Circulating Levels of Ghrelin in Patients With a Rare Disease Associated With Intellectual Disability, and Hyperphagia, and / or Overweight, and / or Obesity
Brief Title: Ghrelin in Patients With a Rare Disease Associated With Intellectual Disability, and Hyperphagia, and/or Overweight, and/or Obesity
Acronym: HOGRID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0176
Record Dates: First submitted 2021-02-16; First posted 2021-02-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Angelman Syndrome; Smith-Magenis Syndrome; X Fragile Syndrome; Epilepsy; Prader-Willi Syndrome
MeSH Terms: conditions — Angelman Syndrome; Smith-Magenis Syndrome; Fragile X Syndrome; Epilepsy; Prader-Willi Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — collection de plasma et cellules sanguines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: acylated and unacylated ghrelin dosages — realization of plasma samples to evaluate of levels of ghrelin and collection of plasma and cells

SUMMARY:
A significantly higher proportion of patients with rare diseases (RD) with intellectual disability (ID), present hyperphagia, overweight or obesity, compared to the general population. Prader-Willi syndrome is the only genetic obesity identified to date associated with hyperghrelinemia, while ghrelin levels are lower than in controls in other situations of obesity.

The aim of the study is to find out whether the levels of ghrelin, which are abnormally high in PWS throughout life, are also high in these RD when people have hyperphagia and/or overweight.

DETAILED DESCRIPTION:
A significantly higher proportion of patients with rare diseases (RD) with intellectual disability (ID), present hyperphagia, overweight or obesity, compared to the general population. Prader-Willi Syndrome (PWS) and related syndromes (PWS-like) represent the most well-known causes of eating disorders with early and severe obesity. Other known RD with ID have been described as being associated with eating disorders with overweight or obesity, which appear later in adolescence : Angelman's syndrome (approximately 40% of patients are overweight or obese, and 32% of children have hyperphagia), Fragile X syndrome (over 30% are obese), Smith-Magenis syndrome (50 to 60% are obese). Prader-Willi syndrome is the only genetic obesity identified to date associated with hyperghrelinemia, while ghrelin levels are lower than in controls in other situations of obesity.

The aim of the study is to find out whether the levels of ghrelin, which are abnormally high in PWS throughout life, are also high in these pathologies when people have hyperphagia and/or overweight.

The study involves a single visit carried out during a routine follow-up in the CRMR, in which the blood sample will allow the dosage of the ghrelin hormon. The visit will also involves a data collection and some questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of the following rare diseases associated with : Angelman syndrome, Smith-Magenis syndrome, X Fragile syndrome, rare diseases of the cerebellum, rare epilepsies, PW-like syndromes or other rare diseases with eating disorders
* Patients aged minimum 3 years and maximum 50 years.
* Patients with overweight (or obesity) and/or hyperphagic behavior.

Exclusion Criteria:

* Administrative problems: impossibility of giving parents or legal guardians informed information ; no coverage by a Social Security scheme.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients infants and adults presenting a rare disease with overweight and hyperphagic behavior
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Levels of ghrelin in blood sample | Day 1
  dosage of ghrelin (pmol /l)

SECONDARY OUTCOMES:
Overeating | Day 1
  Dykens overeating questionnaire
Overeating | Day 1
  eating behavior assessment scale
Behavioral disorder description | Day 1
  CBCL questionnaire for patients under 18 years old
Behavioral disorder description | Day 1
  Developmental Behavior Checklist-Adult questionnaire for patients over 18 years old
Social vulnerability of parents and / or legal guardians | Day 1
  EPICES questionnaire (Assessment of Precariousness and Health Inequalities for the Health Examination Centers).
Family quality of life (for patients under 18) | Day1
  Parental-Developmental Disabilities Quality of Life questionnaire
Burden of parents and / or legal guardians | Day 1
  ZBI questionnaire (Zarit Burden Interview).

CONTACTS AND LOCATIONS:
Overall Officials: Maithé TAUBER, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - Centre N°1 : 40 Centre de Référence PRADORT Pr Tauber - Toulouse Centre N°2 : 22 Centre de Référence PRADORT Pr Poitou Bernert - Paris La Pitié Salpetrière Centre N°3 : 15 Centre de Référence DI de causes rares Dr Heron - Paris La Pitié Salpêtrière Centr, Paris
  - Tauber, Toulouse

IPD SHARING:
Plan to Share IPD: No